CLINICAL TRIAL: NCT07040631
Title: Effect of Hyaluronic Acid on Post-Intubation Sore Throat and Hoarseness in Breast Cancer Surgery: A Randomized Controlled Trial
Brief Title: Hyaluronic Acid for Prevention of Post-Intubation Sore Throat and Hoarseness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 21-2025-006
Record Dates: First submitted 2025-05-20; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Postoperative Sore Throat, Cough, Hoarseness; Endotracheal Intubation; General Anesthesia
Keywords: Postoperative Sore Throat; Hyaluronic Acid; Lubricating Gel; Endotracheal Intubation; hoarseness; breast cancer surgery; randomized controlled trial
MeSH Terms: conditions — Breast Neoplasms; Cough; Hoarseness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endogra Gel Group (Experimental): Participants will receive general anesthesia for breast cancer surgery. Endotra Gel, a hyaluronic acid-based gel, will be applied evenly on the surface of the endotracheal tube cuff prior to intubation.
  Interventions: Device: Endotra Gel
- No Gel Group (No Intervention): Participants will receive standard care for endotracheal intubation under general anesthesia without application of any gel or lubricant to the endotracheal tube.

INTERVENTIONS:
Device: Endotra Gel — Endotra Gel is a hyaluronic acid-based, water-soluble wound dressing gel approved by the Korean Ministry of Food and Drug Safety. In this study, it is applied to the cuff of the endotracheal tube before intubation to evaluate its effect on reducing postoperative sore throat and hoarseness.
  Arms: Endogra Gel Group

SUMMARY:
The goal of this clinical trial is to find out whether applying Endotra Gel, a hyaluronic acid-based gel, to the endotracheal tube can help reduce sore throat and hoarseness after surgery.

These symptoms are common after general anesthesia when a endotracheal tube is placed into the trachea. They can cause discomfort and affect patient recovery.

The main questions this study aims to answer are:

* Does Endotra Gel reduce the chance of having a sore throat after surgery?
* Does it help improve hoarseness or coughing after surgery?

Participants in this study will:

* Undergo general anesthesia for breast cancer surgery
* Be randomly assigned to one of two groups:

  * One group will receive Endotra Gel applied to the endotracheal tube before intubation
  * The other group will have standard care with no gel
* Be monitored for sore throat, hoarseness, and coughing right after surgery and on the day after surgery
* Answer questions about their symptoms and satisfaction with their recovery The results will help researchers learn whether using Endotra Gel during intubation can improve patient comfort and reduce airway irritation after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 to 80 years
* Scheduled to undergo breast cancer surgery under general anesthesia with endotracheal intubation
* American Society of Anesthesiologists (ASA) physical status I to III

Exclusion Criteria:

* Mallampati classification of III or higher
* Recent upper respiratory infection or symptoms of upper airway infection
* Pre-existing laryngeal disease or chronic respiratory conditions (e.g., asthma, chronic bronchitis)
* Current use of systemic steroids
* Refusal to provide informed consent
* Determined to be unsuitable for study participation by the investigator

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Postoperative Sore Throat | Up to 1 hour after extubation at PACU
  Postoperative sore throat (POST) will be assessed using a standardized 4-point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe) through direct patient interview. Assessment will be performed by blinded outcome assessors.

SECONDARY OUTCOMES:
Incidence and Severity of Postoperative Hoarseness | Up to 1 hour after extubation at PACU and on postoperative day 1 (within 24 hours after surgery)
  Hoarseness will be evaluated using a 4-point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe) through patient interview. Evaluation will be performed by blinded assessors.
Incidence and Severity of Postoperative Cough | Up to 1 hour after extubation at PACU and on postoperative day 1 (within 24 hours after surgery)
  Postoperative cough will be assessed on a 4-point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe) through direct questioning. Evaluation will be conducted by blinded assessors.
Patient Satisfaction with Intubation Experience | On postoperative day 1 (within 24 hours after surgery)
  Patient satisfaction regarding intubation-related discomfort will be evaluated using two structured questions:
  "Postoperative discomfort related to intubation interfered with daily life."
  "Overall, I am satisfied with the intubation experience."
  Each item will be rated on a 5-point Likert scale:
  1 = Strongly agree, 2 = Agree, 3 = Neutral, 4 = Disagree, 5 = Strongly disagree.
  Responses will be collected on postoperative day 1 and analyzed as ordinal variables.